CLINICAL TRIAL: NCT05029739
Title: An Interactive E-health Intervention to Promote Walking Capacity and Life-style Changes in Peripheral Artery Disease (iPAD)
Brief Title: An E-health Intervention for Patients With Peripheral Artery Disease
Acronym: I-PAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other); Karlstad Central Hospital (Other); Jonkoping County Hospital (Other); Sidekick Health (Industry)
Responsible Party: Principal Investigator, Joakim Nordanstig, Associate Professor of Vascular Surgery, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-PAD
Record Dates: First submitted 2021-08-17; First posted 2021-09-01 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Intermittent Claudication
Keywords: Peripheral Artery Disease; E-intervention; Best medical therapy
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized open blinded end-point (PROBE)
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded for group assignment at the 12 weeks and 12 month follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-intervention group (Experimental): Participants will be instructed to download a life-style-changing mobile app to which they will have access for 12 weeks. After the first week of the program, participants who smoke will be offered to incorporate smoking cessation support into their PAD program. These changes are minor and not intended to divide the intervention group in two but instead to personalize the study experience. The program aims to empower positive lifestyle change by gamification, altruistic rewards, and engaging content with relevant tasks or missions to be completed. Beyond this, all patients in the interventional arm will also receive standard of care as defined below for the control arm.
  Interventions: Device: A PAD-specific smartphone application (e-intervention) developed for patients with Peripheral Artery Disease
- Standard of care - control group. (Active Comparator): All patients in the control arm will receive best medical therapy including start or optimization of secondary preventive pharmacotherapy, smoking cessation advise and advise on modifiable risk factors. The control arm will also receive an information leaflet about relevant lifestyle modifications for PAD. After the baseline measurements and data collection, there will be no scheduled visits to a health care provider until week 12.
  Interventions: Device: A PAD-specific smartphone application (e-intervention) developed for patients with Peripheral Artery Disease

INTERVENTIONS:
Device: A PAD-specific smartphone application (e-intervention) developed for patients with Peripheral Artery Disease — See description of the e-intervention group as above.

SUMMARY:
The specific study aim is to determine whether a 12-week digitally delivered behavior change intervention for patients with peripheral artery disease increases walking ability, reduces smoking, improves quality of life and improves medication adherence. The primary and secondary endpoints will primarily be captured at a 12 weeks follow-up visit, but a follow-up visit after 12 months is also planned; to assess longer term effect on outcomes and healthcare cost.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a highly prevalent atherosclerotic syndrome with an estimated global population burden of ~200 million people. PAD patients are at heightened risk for adverse cardiovascular- and limb events and impaired quality of life. Cigarette smoking is the most important modifiable risk factor. Patients with PAD who smoke have higher disease progression rates, greater risk of complications, poor post-procedural outcomes, compromised functional status, and increased hospitalizations.

A significant goal of PAD treatment includes risk factor modification and prevention of cardiovascular events. Guideline-directed therapy includes cardioprotective pharmacotherapies, and lifestyle modification. Nevertheless, adherence to pharmacologic and lifestyle recommendations in PAD is uncertain. Effective non-pharmacologic therapies for PAD also exist, including smoking cessation, exercise support, and diet counseling. However, limited data is available on mobile applications offering digitally delivered lifestyle change support, including a structured exercise program and smoking cessation support. This study aims to digitally provide lifestyle change support, including a structured and PAD-focused lifestyle program and smoking cessation support via a mobile platform (Sidekick Health) with the primary aim to increase patients' walking ability and secondary aims to reduce smoking and improve medication adherence.

Hypotheses

1. At the end of the 12 weeks, the interventional arm will reach a clinically meaningful change in walking ability, as compared to controls, measured by a change in the 6-MWT at twelve-week, and 12 months; the minimal clinically important difference (MCID) is defined as +12m.
2. At the end of the 12 weeks, ≥15% interventional treatment arm participants will give up smoking or have significantly reduced their daily smoking compared to less than <10% in the control arm.
3. At the end of the 12 weeks, ≥50% of interventional treatment arm participants will improve their medication adherence from pre- until post-intervention as compared to <30% in the control arm.
4. Healthcare cost will be reduced at 12 month follow-up in the intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Adults with confirmed PAD referred to a vascular surgery unit for evaluation and treatment, currently on best medical treatment and own/have access to a mobile smartphone
* Stable PAD disease and limb symptoms during the last 3 months.
* PAD is the activity-limiting disease
* Abnormal resting ankle-brachial index (ABI) (≤0.90), falsely elevated ABI above 1.3 or a 30% post-exercise ABI reduction.

Exclusion Criteria:

* Critical limb ischemia, prior amputation, or other diseases/ impairment that limit the walking ability and the 6-minute walk test's proper conduct
* Cognitive impairment
* Prior revascularization less than one year ago
* A planned revascularization procedure during the upcoming 12 months (known at baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test. | 12 weeks and 12 months
  Change in objectively measured (pain-free and maximal) walking capacity (as measured with the 6-Minute Walk Distance Test) from baseline to 12 weeks and 12 months

SECONDARY OUTCOMES:
Smoking status | 12 weeks and 12 months
  Change in patients´ daily smoking patterns from pre to post-intervention and at 12-months. This outcome will be measured through a carbon mononoxide exhalor test and by patient-reported daily frequency of cigarettes smoked at baseline, 12 weeks and 12 months
Increased readiness to quit smoking. | 12 weeks and 12 months
  This outcome will be measured through the smoking 'Readiness to quit' questionnaire (The Contemplation Ladder) at baseline, 12 weeks and 12 months.
Medication adherence improvement | 12 weeks and 12 months
  To determine patients' adherence to their medications after the usage of the smartphone application as compared to standard of care. This secondary outcome will be measured through a questionnaire; Morisky Medication Adherence Scale, MMAS-8 at baseline, 12 weeks and 12 months.
Disease-specific health-related quality of life. | 12 weeks and 12 months
  Health related quality of life; measured by the disease-specific questionnaire VascuQoL-6 at baseline, 12 weeks and 12 months.
Comparing outcomes to health literacy | 12 weeks and 12 months
  Comparing outcomes to health literacy measured through a questionnaire; HLS-EU-Q16 at baseline.
Quality Adjusted Life Years (QALYs) | 12 months
  Calculated based on recorded accumulated costs and registered EQ5D-5L outcomes
Change in self-assessed stress levels | 12 weeks
  Self-reported ordinal scale ranging from 0 to 10
Change in self-assessed sleep quality levels | 12 weeks
  Self-reported ordinal scale ranging from 0 to 10
Change in self-assessed energy levels | 12 weeks
  Self-reported ordinal scale ranging from 0 to 10
Change in free living physical activity | 12 Weeks
  Measured as total step count per day

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Nordanstig, MD,PhD, Principal Investigator — Institute of Medicine at the Sahlgrenska Academy, University of Gothenburg, Sweden.
Locations (5):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Jönköping Central Hospital, Jönköping
  - Karlstad Central Hospital, Karlstad
  - Skane University Hospital, Malmo
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No
Anonymized IPD may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT05029739/Prot_SAP_000.pdf